CLINICAL TRIAL: NCT02324426
Title: Central Nervous System Uptake of Intranasal Glutathione in Parkinson's Disease
Brief Title: CNS Uptake of Intranasal Glutathione
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Laurie Mischley, Project Appointment, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48273-A
Record Dates: First submitted 2014-12-04; First posted 2014-12-24 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Reduced Glutathione; CNS; Glutathione; Uptake; Intranasal; (in)GSH
MeSH Terms: conditions — Parkinson Disease | interventions — Glutathione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced Glutathione (Experimental): The study medication is packaged in sterile 1 ml pre-filled syringes, each containing 200 mg/ ml of reduced glutathione (GSH), which will be delivered intranasally.
  Interventions: Drug: Reduced Glutathione

INTERVENTIONS:
Drug: Reduced Glutathione — 200 mg GSH delivered in 1 cc sterile saline using a syringe with a Mucosal Atomization Device (MAD) tip.
  Other Names: (in)GSH

SUMMARY:
Excessive free radical formation and depletion of the brain's primary antioxidant, glutathione, are established components of Parkinson's disease (PD) pathophysiology. While there is rationale for the therapeutic use of reduced glutathione (GSH) in PD, and even some preliminary evidence to suggest the use of GSH can lead to symptomatic improvement, obstacles surrounding currently employed delivery methods have hindered the clinical utility of this therapy. Intranasal GSH, (in)GSH, is a novel method of glutathione augmentation. The aim of this study is to evaluate whether 200 mg of (in)GSH results in measurable changes in brain glutathione concentrations, as measured by magnetic resonance spectroscopy (MRS) in 15 individuals with PD.

DETAILED DESCRIPTION:
Objectives

Primary Aim: To determine whether intranasal reduced glutathione, (in)GSH, is capable of augmenting CNS glutathione levels.

Hypothesis: Mean MRS glutathione concentration will rise from baseline following administration of 1 cc 200 mg/ml (in)GSH.

Design and Outcomes:

This pilot study seeks to obtain baseline data regarding the feasibility of MRS to detect a change in CNS glutathione concentration following administration of 200 mg (in)GSH. CNS glutathione levels will be measured using magnetic resonance spectroscopy (MRS), with the putamen as the region of interest. Baseline brain GSH concentrations will be measured by MRS at approximately the same time each day in all individuals before and after administration of study medication.

Outcome Measure: Describe the change in mean GSH concentration following administration of (in)GSH. The data analysis will be ipsative- results will be reported as percent change from the individual's own baseline GSH concentration.

Interventions and Duration:

If a participant communicates he/she understands the study, meets inclusion criteria, and provides informed consent, individuals will be scheduled for a single visit at the University of Washington for MR imaging (MRI), clinical evaluation, and blood draw. (~ 3 hours). Participants will be asked to be optimally medicated at the time of study visit, to the best of their ability.

Sample Size and Population:

This is a proof-of-concept pilot trial. Based on the data from the single test subject, a sample size of 15 would provide 80% power to detect an increase in CNS glutathione concentrations between pre- and post- administration values, if we are willing to accept an alpha value of 0.2.

1.1 Primary Aims

Primary Aim: To determine whether intranasal reduced glutathione, (in)GSH, is capable of augmenting CNS glutathione concentration. (Region of Interest: putamen)

Hypothesis: Mean MRS glutathione concentration will rise from baseline approximately 15 minutes following administration of 200 mg/ml (in)GSH in 1 cc saline.

1.2 Secondary Objectives

Hypothesis: Baseline CNS glutathione concentrations and RBC glutathione concentrations will be correlated.

1. To determine whether brain MRS [glutathione] and red blood cell (RBC) glutathione levels are correlated.

Outcome: A ROC curve will be drawn between mean brain [glutathione] and RBC total glutathione.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Ability to attend a 3 hour study visit in Seattle, WA.
* Ability to read and speak English.
* Have three or more of the required positive criteria for PD from Step 3 of the UK Brain Bank Diagnostic Criteria for Parkinson's Disease.
* A modified Hoehn & Yahr Stage 2-3. (bilateral disease, not severely disabled.)

Exclusion Criteria:

* Any contra-indication to magnetic resonance imaging, including pacemaker, pacemaker wires, aneurysm clip, or any electronic implant, weight over 136 kg (300 lb), metal embedded in soft tissue or in the eye, prosthetic eye, claustrophobia, substance abuse, use of recreational drugs, pregnancy, or other medical contraindications.
* A history of epilepsy, stroke, brain surgery, or structural brain disease.
* The presence of other serious illnesses (discretion of study clinician, e.g. concurrent cancer treatment.)
* Pregnant.
* A history of sulfur sensitivity, e.g. reaction N-acetylcysteine, MSM, SAMe.
* A recent history of asthma.
* Supplementation with glutathione (oral, intravenous, intranasal, or nebulized) or the glutathione precursor, N-acetylcysteine, for six months prior to baseline study visit.
* History of sensitivity to sulfur containing medications/ supplements, i.e. NAC, MSM.
* Current drug or alcohol use or dependence.
* Inability/unwillingness to provide informed consent. (e.g. diagnosis of dementia, confusion about study goals or participation.)
* Acute infection (e.g. upper respiratory, dermal) in the previous 30 days.
* Diagnosis of any mental illness, ever. (Mental illness has been associated with glutathione depletion.)
* Diagnosis of any chronic disease, ever. (e.g. Hep C, autoimmune disease, etc.)
* Head tremor or head dyskinesia that cannot be comfortably controlled for 90 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The concentration of metabolites before and after (in)GSH will be compared (change in mean GSH concentration) | 15 minutes after administration
  Describe the change in mean GSH concentration following administration of (in)GSH. The data analysis will be ipsative- results will be reported as percent change from the individual's own baseline GSH concentration.

SECONDARY OUTCOMES:
A ROC curve will be generated to compare MRS [glutathione] to peripheral measures of RBC glutathione. | 15 minutes after administration

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Conley, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Coyle JT, Puttfarcken P. Oxidative stress, glutamate, and neurodegenerative disorders. Science. 1993 Oct 29;262(5134):689-95. doi: 10.1126/science.7901908.
- [Background] Mischley, L. Glutathione Deficiency in Parkinson's Disease: Intranasal Administration as a Method of Augmentation. Journal of Orthomolecular Medicine 26(1):32-36, 2011.
- [Background] Bains JS, Shaw CA. Neurodegenerative disorders in humans: the role of glutathione in oxidative stress-mediated neuronal death. Brain Res Brain Res Rev. 1997 Dec;25(3):335-58. doi: 10.1016/s0165-0173(97)00045-3. PMID 9495562
- [Background] Cacciatore I, Baldassarre L, Fornasari E, Mollica A, Pinnen F. Recent advances in the treatment of neurodegenerative diseases based on GSH delivery systems. Oxid Med Cell Longev. 2012;2012:240146. doi: 10.1155/2012/240146. Epub 2012 Jun 3. PMID 22701755
- [Background] Shils ME OJ, Shike, Moshe. Evolution of Knowledge of Essential Nutrients: Conditional Essentiality. Modern Nutrition in Health and Disease. Philadelphia: Lippincott Williams & Wilkins; 2006.
- [Background] Mullins PG, McGonigle DJ, O'Gorman RL, Puts NA, Vidyasagar R, Evans CJ; Cardiff Symposium on MRS of GABA; Edden RA. Current practice in the use of MEGA-PRESS spectroscopy for the detection of GABA. Neuroimage. 2014 Feb 1;86:43-52. doi: 10.1016/j.neuroimage.2012.12.004. Epub 2012 Dec 13. PMID 23246994
- [Background] Maher P. The effects of stress and aging on glutathione metabolism. Ageing Res Rev. 2005 May;4(2):288-314. doi: 10.1016/j.arr.2005.02.005. PMID 15936251
- [Result] Pocernich CB, Cardin AL, Racine CL, Lauderback CM, Butterfield DA. Glutathione elevation and its protective role in acrolein-induced protein damage in synaptosomal membranes: relevance to brain lipid peroxidation in neurodegenerative disease. Neurochem Int. 2001 Aug;39(2):141-9. doi: 10.1016/s0197-0186(01)00012-2. PMID 11408093
- [Result] Sian J, Dexter DT, Lees AJ, Daniel S, Agid Y, Javoy-Agid F, Jenner P, Marsden CD. Alterations in glutathione levels in Parkinson's disease and other neurodegenerative disorders affecting basal ganglia. Ann Neurol. 1994 Sep;36(3):348-55. doi: 10.1002/ana.410360305. PMID 8080242
- [Result] Sofic E, Lange KW, Jellinger K, Riederer P. Reduced and oxidized glutathione in the substantia nigra of patients with Parkinson's disease. Neurosci Lett. 1992 Aug 17;142(2):128-30. doi: 10.1016/0304-3940(92)90355-b. PMID 1454205
- [Result] Sechi G, Deledda MG, Bua G, Satta WM, Deiana GA, Pes GM, Rosati G. Reduced intravenous glutathione in the treatment of early Parkinson's disease. Prog Neuropsychopharmacol Biol Psychiatry. 1996 Oct;20(7):1159-70. doi: 10.1016/s0278-5846(96)00103-0. PMID 8938817
- [Result] Mischley LK SL, Samii A, Pollisar N, Lau R, Leverenz J, . Phase I Study of Intranasal Glutathione in Parkinson's Disease. Seattle: Bastyr University Research Instittue; 2013.
- [Result] Lee M, Cho T, Jantaratnotai N, Wang YT, McGeer E, McGeer PL. Depletion of GSH in glial cells induces neurotoxicity: relevance to aging and degenerative neurological diseases. FASEB J. 2010 Jul;24(7):2533-45. doi: 10.1096/fj.09-149997. Epub 2010 Mar 12. PMID 20228251
- [Result] Pearce RK, Owen A, Daniel S, Jenner P, Marsden CD. Alterations in the distribution of glutathione in the substantia nigra in Parkinson's disease. J Neural Transm (Vienna). 1997;104(6-7):661-77. doi: 10.1007/BF01291884. PMID 9444566
- [Result] DelleDonne A, Klos KJ, Fujishiro H, Ahmed Z, Parisi JE, Josephs KA, Frigerio R, Burnett M, Wszolek ZK, Uitti RJ, Ahlskog JE, Dickson DW. Incidental Lewy body disease and preclinical Parkinson disease. Arch Neurol. 2008 Aug;65(8):1074-80. doi: 10.1001/archneur.65.8.1074. PMID 18695057
- [Result] Witschi A, Reddy S, Stofer B, Lauterburg BH. The systemic availability of oral glutathione. Eur J Clin Pharmacol. 1992;43(6):667-9. doi: 10.1007/BF02284971. PMID 1362956
- [Result] Hauser RA, Lyons KE, McClain T, Carter S, Perlmutter D. Randomized, double-blind, pilot evaluation of intravenous glutathione in Parkinson's disease. Mov Disord. 2009 May 15;24(7):979-83. doi: 10.1002/mds.22401. PMID 19230029
- [Result] Emir UE, Raatz S, McPherson S, Hodges JS, Torkelson C, Tawfik P, White T, Terpstra M. Noninvasive quantification of ascorbate and glutathione concentration in the elderly human brain. NMR Biomed. 2011 Aug;24(7):888-94. doi: 10.1002/nbm.1646. Epub 2011 Jan 12. PMID 21834011
- [Result] Groger A, Chadzynski G, Godau J, Berg D, Klose U. Three-dimensional magnetic resonance spectroscopic imaging in the substantia nigra of healthy controls and patients with Parkinson's disease. Eur Radiol. 2011 Sep;21(9):1962-9. doi: 10.1007/s00330-011-2123-5. Epub 2011 Apr 12. PMID 21484351
- [Result] Emir UE, Deelchand D, Henry PG, Terpstra M. Noninvasive quantification of T2 and concentrations of ascorbate and glutathione in the human brain from the same double-edited spectra. NMR Biomed. 2011 Apr;24(3):263-9. doi: 10.1002/nbm.1583. Epub 2010 Oct 6. PMID 20925125
- [Result] Sekhar RV, Patel SG, Guthikonda AP, Reid M, Balasubramanyam A, Taffet GE, Jahoor F. Deficient synthesis of glutathione underlies oxidative stress in aging and can be corrected by dietary cysteine and glycine supplementation. Am J Clin Nutr. 2011 Sep;94(3):847-53. doi: 10.3945/ajcn.110.003483. Epub 2011 Jul 27. PMID 21795440
- [Result] Holmay MJ, Terpstra M, Coles LD, Mishra U, Ahlskog M, Oz G, Cloyd JC, Tuite PJ. N-Acetylcysteine boosts brain and blood glutathione in Gaucher and Parkinson diseases. Clin Neuropharmacol. 2013 Jul-Aug;36(4):103-6. doi: 10.1097/WNF.0b013e31829ae713. PMID 23860343
- [Result] Mischley LK, Vespignani MF, Finnell JS. Safety survey of intranasal glutathione. J Altern Complement Med. 2013 May;19(5):459-63. doi: 10.1089/acm.2011.0673. Epub 2012 Dec 16. PMID 23240940